CLINICAL TRIAL: NCT06749730
Title: A Prospective, Single Arm Study of Adebrelimab Combined with Apatinib and Gemcitabine and Cisplatin (GP) First-line Treatment for Unresectable Biliary Tract Carcinoma
Brief Title: Adebrelimab Combined with Apatinib and Gemcitabine and Cisplatin (GP) First-line Treatment for Unresectable Biliary Tract Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Ying Liu, Deputy Chief Physician, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTC-II-001
Record Dates: First submitted 2024-07-11; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-07

CONDITIONS: Unresectable Biliary Tract Carcinoma
MeSH Terms: interventions — apatinib; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- adebrelimab combined with apatinib and gemcitabine and cisplatin (Experimental)
  Interventions: Drug: Adebrelimab; Drug: Apatinib; Drug: gemcitabine and cisplatin

INTERVENTIONS:
Drug: Adebrelimab — adepelizumab ,1200mg, q3w
Drug: Apatinib — apatinib，250mg，QD
Drug: gemcitabine and cisplatin — cisplatin 25mg/m2，gemcitabine 1000mg/m2 d1,d8，q3w

SUMMARY:
This study is designed to combine anti-angiogenic drugs on the basis of PD-L1+ gemcitabine/cisplatin, hoping to further improve the curative effect of advanced BTC treatment and provide more choices for first-line treatment of BTC in China.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age range from 18 to 80 years old, regardless of gender;
* 2.Histologically confirmed, unresectable advanced or metastatic BTC including cholangiocarcinoma (intrahepatic or extrahepatic), gallbladder carcinoma.
* 3. Patients who have not received systematic treatment for BTC in the past .
* 4.At least one measurable lesion (according to RECIST v1.1 requirements).
* 5.ECOG PS: 0-1 points;
* 6.Expected survival time ≥ 12 weeks;
* 7. The main organs are functioning normally and meet the following requirements White blood cell count ≥ 3.0× 10 9/L; Hb ≥ 90 g/l; Absolute neutrophil count ≥ 1.5× 10 9/L; Platelet count ≥ 100× 10 9/L; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤ 2.5 times the upper limit of normal limit (ULN); Total bilirubin ≤ 2 times of ≤ULN; Serum creatinine ≤ 1.5 times of ≤ULN; Albumin ≥ 30 g/l;
* 8. Women of childbearing age must undergo a pregnancy test (serum or urine) with a negative result within 14 days prior to enrollment, and voluntarily use appropriate methods of contraception during observation and within 8 weeks after the last administration of study medication; For males, surgical sterilization should be performed, or appropriate methods of contraception should be agreed upon during observation and within 8 weeks after the last administration of study medication;
* 9. The subjects voluntarily joined this study, signed an informed consent form, and cooperated with follow-up.

Exclusion Criteria:

* 1. Histologically diagnosed as neuroendocrine carcinoma;
* 2. People who are allergic to adebelizumab, apatinib, gemcitabine, cisplatin or their auxiliary materials;
* 3. Systemic treatment in the past;
* 4. Pleural effusion, pericardial effusion or ascites accompanied by clinical symptoms and judged by the researcher to require frequent drainage;
* 5. History of organ transplantation (including autologous bone marrow transplantation and peripheral stem cell transplantation);
* 6. Active or uncontrollable serious infection (≥ CTCAE grade 5.02 infection), including but not limited to hospitalization due to infection complications, bacteremia or severe pneumonia, and unexplained fever > 38.5℃ before the first administration;
* 7. Liver cirrhosis and active hepatitis; Hepatitis B reference: HBsAg positive, and HBV DNA exceeds the upper limit of normal value (1000 copies /ml or 500 IU/ml); Patients with hepatitis B virus (HBV) infection or cured HBV infection in the past (defined as the existence of hepatitis B core antibody [HBcAb] and the absence of HBsAg, and those with normal HBV DNA value during the screening period can be included; Hepatitis C reference: HCV antibody is positive, and the detection value of HCV virus titer exceeds the upper limit of normal value /HCV RNA or HCV Ab detection indicates acute and chronic infection;
* 8. Those who have a history of psychotropic drug abuse and cannot quit or have mental disorders;
* 9.Within 5 years, the subject has other malignant tumors in the past or at the same time and needs active treatment (except for fully treated basal cell or squamous cell skin cancer, cervical carcinoma in situ and breast cancer in situ, if the estimated 5-year survival rate is more than 90%);
* 10. There is an uncorrectable coagulation disorder;
* 11. Severe liver diseases (such as liver cirrhosis), kidney diseases, respiratory diseases, uncontrollable diabetes or other types of systemic diseases.
* 12. Patients whose imaging shows that the tumor has invaded important blood vessels or who are judged by the researchers to be very likely to invade important blood vessels and cause fatal bleeding during the follow-up study;
* 13. Active autoimmune disease or immunodeficiency, or the following medical history, including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, rheumatoid arthritis, inflammatory bowel disease, hypophysitis, vasculitis, nephritis, etc.) shall not be included. The following exceptions are made: patients with a history of autoimmune hypothyroidism but receiving thyroid hormone replacement therapy can be included in the study. Patients with type 1 diabetes whose blood sugar has been controlled after insulin administration can participate in this study.
* 14, Within 14 days prior to signing the informed consent form, use immunosuppressive agents or systemic hormone therapy to achieve immunosuppressive effects (dose>10mg/day prednisone or other therapeutic hormones)
* 15.Arterial/venous thrombosis events occurred within 6 months before the first administration, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral embolism, etc.), deep venous thrombosis and pulmonary embolism;
* 16.The researcher judges digestive tract diseases or conditions that may affect drug absorption, including but not limited to active gastric and duodenal ulcers, ulcerative colitis or active bleeding of unresectable digestive tract tumors, or other conditions that may cause gastrointestinal bleeding or perforation as judged by the researcher, with various factors that affect oral drugs (such as inability to swallow, gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc.);
* 17.Individuals with hypertension who cannot be reduced to the normal range after antihypertensive drug treatment (systolic blood pressure ≥ 150mmHg or diastolic blood pressure ≥ 100mmHg)
* 18.Surgery (except biopsy) was performed within 28 days before being enrolled in this study, or the surgical incision was not completely healed;
* 19.Have received any other experimental drug treatment or participated in other intervention research within 4 weeks before signing the informed consent form;
* 20.Pregnant (pregnancy test positive before medication) or breast-feeding women;
* 21.According to the researcher's judgment, that is not suitable for patients in the group;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | From first dose of study intervention until disease progression or death (whichever occurs first), up to approximately 6 months after the last subject enrolled
  Progression-free Survival (PFS) is defined as the time from randomization to the first documented radiographic disease progression or death due to any cause, whichever occurs first, assessed by the Investigator per RECIST Version 1.1.

SECONDARY OUTCOMES:
Overall Survival(OS) | From first dose of study intervention until death, at least 12 months after the last subject enrolled
  Overall Survival(OS) is defined as the time from the date of the first dose of study intervention until death due to any cause. The measures of interest are median Overall Survival(OS) and Overall Survival at 12 months(OS12).
Objective Response Rate (ORR) | From first dose of study intervention until disease progression or death (whichever occurs first), up to approximately 3 months after the last subject enrolled
  Objective Response Rate (ORR) is defined as the proportion of participants who achieved a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR), assessed by BICR per RECIST Version 1.1.
Duration of Response(DOR) | From first dose of study intervention until disease progression or death (whichever occurs first), up to approximately 6 months after the last subject enrolled
  Duration of Response(DOR) is defined as the time from the date of first documented response until the date of documented progression per RECIST 1.1 as assessed by the investigator or death due to any cause.
Incidence of treatment-emergent adverse events(AEs) | From first dose of study intervention until 90 days after last dose or death (whichever occurs first)
  Incidence of treatment-emergent adverse events(AEs), including possible related adverse events(PRAEs), adverse event of special interests(AESIs), immune-mediated adverse events(imAEs), and serious adverse events(SAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Ying Liu, MD, Principal Investigator — Study Principal Investigator Henan Cancer Hospital
Locations (1):
- HeNan, Zhengzhou, China